CLINICAL TRIAL: NCT06990607
Title: Pars Plana Vitrectomy With Silicone Oil Versus Pars Plana Vitrectomy Alone in the Management of Postoperative Endophthalmitis
Brief Title: Compare PPV With and Without Silicone Oil in Managing Postoperative Endophthalmitis
Acronym: Endopthalmitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endophthalmitis and silicone
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Endophthalmitis Following Cataract Surgery
Keywords: Postoperative endophthalmitis; pars plana vitrectomy; silicone oil
MeSH Terms: interventions — Silicone Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Pars plana Vitrectomy Alone
  Interventions: Procedure: Pars plana Vitrectomy
- Group II (Active Comparator): Pars plana Vitrectomy with Silicone Oil
  Interventions: Procedure: Pars plana Vitrectomy; Procedure: Silicone Oil

INTERVENTIONS:
Procedure: Pars plana Vitrectomy — Pars plana Vitrectomy using 23 Gauge
Procedure: Silicone Oil — Silicone Oil injection after PPV
  Arms: Group II

SUMMARY:
Comparing PPV with and without silicone oil in managing postoperative endophthalmitis

DETAILED DESCRIPTION:
The objective of this study is to compare the outcomes of PPV with silicone oil tamponade to PPV alone in patients with postoperative endophthalmitis by assessing visual acuity, and postoperative complications such as rhegmatogenous retinal detachment (RRD).

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years) presenting with clinical manifestations of endophthalmitis after cataract surgery

Exclusion Criteria:

* patients with concurrent ocular or systemic conditions that could potentially confound study outcomes, such as active retinal diseases unrelated to endophthalmitis
* pre-existing poor visual prognosis due to conditions like advanced glaucoma or macular degeneration, or prior ocular surgery affecting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
visual acuity, with best-corrected visual acuity (BCVA) recorded using LogMAR | 1, 2, 4, and 12 weeks postoperatively
  log-MAR value (log of the minimum angle of resolution). Normal visual acuity for most adults is approximately -0.1 on this scale, which is equivalent to 20/16 on a Snellen visual acuity chart.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Cairo Governorate, Egypt